CLINICAL TRIAL: NCT00698659
Title: A Study of the Pharmacodynamic Effects of Anti-Vascular Endothelial Growth
Brief Title: Pharmacodynamic Effects of Anti-Vascular Endothelial Growth Factor Therapy in Patients With Advanced Malignancies
Status: Terminated | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: MC2/15/07
Record Dates: First submitted 2008-06-15; First posted 2008-06-17 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2012-04

CONDITIONS: Hypertension; Proteinuria
MeSH Terms: conditions — Hypertension; Proteinuria

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients on anti-VEGF therapy: This study aims to assess the pharmacodynamic effects of anti-VEGF therapy. The following groups of patients will be approached:
  Those who are starting on anti-VEGF therapy (such as but not limited to bevacizumab, sunitinib, and sorafenib) as part of routine clinical management or on clinical studies
  All patients must be aged aged ≥ 21 years All patients must have a signed written informed consent prior to study enrollment. A separate consent will be obtained from patients already involved in a clinical study using anti-VEGF treatment.
  Patients with a known allergy to intravenous contrast used in fluorescein and indocyanine green angiography will be exempt from these investigations but will undergo other study assessments.

SUMMARY:
1. To determine the effect of anti-vascular endothelial growth factor (VEGF) on endothelial function and on retinal microvasculature
2. To determine endothelial dysfunction as a marker of early response and as an indicator for the development of hypertension and proteinuria in patients treated with anti-VEGF agents
3. To characterize the effect of anti-VEGF therapy on the pulmonary function of patients with malignancy (primary or secondary) involving the lung

DETAILED DESCRIPTION:
The well-established role of vascular endothelial growth factor (VEGF) in carcinogenesis and tumor angiogenesis has led to the development of agents that target this pathway. Anti-VEGF agents the VEGF monoclonal antibody bevacizumab, and the small molecule VEGF receptor tyrosine kinase inhibitors. Angiogenic factors play a key role in the maintenance of lung integrity and normal endothelial function. Endothelial dysfunction has been implicated in hypertension, proteinuria and retinopathy. One of the major issues of anti-VEGF agents is its long-term toxicity especially taking into account the lack of adequate knowledge in this area and the possibility of prolonged periods of therapy in non-progressing patients. Hypertension and proteinuria are commonly seen in patients treated with anti-VEGF agents. In addition, we have also observed in a relatively high frequency of pulmonary air-filled lesions in patients with malignancy in the lung treated with an anti-VEGF agent. Objectives of this exploratory study are to 1) determine the effect of anti-vascular endothelial growth factor (VEGF) on endothelial function 2) determine endothelial dysfunction as a marker of early response and as an indicator for the development of hypertension and proteinuria 3) characterize the effect of anti-VEGF therapy on the pulmonary function of patients with malignancy (primary or secondary) involving the lung in patients treated with anti-VEGF agents. Pharmacodynamic endpoints to be assessed are: blood pressure, brachial artery reactivity, retinal microvessels, microalbuminuria and proteinuria, pulmonary function, assess the effects of anti-VEGF therapy by assessing brachial artery reactivity, retinal vasculature and pulmonary function in a subset of patients receiving anti-VEGF therapy. The development of markers of endothelial dysfunction may result in the early identification of patients who are non-responders or develop toxicity from anti-VEGF treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are receiving single agent anti-VEGF therapy
* Signed written informed consent.
* Patients with measurable pulmonary malignancy (primary or metastatic) as determined by RECIST will undergo assessment of pulmonary function.
* Patients with a known allergy to intravenous contrast used in fluorescein and indocyanine green angiography will be exempt from these investigations but will undergo other study assessments

Exclusion Criteria:

* none

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those who are starting on anti-VEGF therapy (such as but not limited to bevacizumab, sunitinib, and sorafenib) as part of routine clinical management
Sampling Method: Non-Probability Sample
Dates: Start 2007-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Effect of VEGF on endothelial function and on retinal microvasculature and the pulmonary function of patients with malignancy (primary or secondary) involving the lung. | until 4 weeks after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ross Andrew Soo, MBBS, MRCP, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Kasahara Y, Tuder RM, Taraseviciene-Stewart L, Le Cras TD, Abman S, Hirth PK, Waltenberger J, Voelkel NF. Inhibition of VEGF receptors causes lung cell apoptosis and emphysema. J Clin Invest. 2000 Dec;106(11):1311-9. doi: 10.1172/JCI10259. PMID 11104784
- [Background] Veronese ML, Mosenkis A, Flaherty KT, Gallagher M, Stevenson JP, Townsend RR, O'Dwyer PJ. Mechanisms of hypertension associated with BAY 43-9006. J Clin Oncol. 2006 Mar 20;24(9):1363-9. doi: 10.1200/JCO.2005.02.0503. Epub 2006 Jan 30. PMID 16446323